CLINICAL TRIAL: NCT01223131
Title: A 24-week, Randomized, Open-label, Parallel Group, Multicenter Comparison of Lantus® (Insulin Glargine) Given Once Daily Versus Neutral Protamine Hagedorn (NPH) Insulin in Children With Type 1 Diabetes Mellitus Aged at Least 6 Years to Less Than 18 Years
Brief Title: Efficacy and Safety of Insulin Glargine Versus. Neutral Protamine Hagedorn (NPH) Insulin in Children With Type 1 Diabetes Above 6 Years Old.
Acronym: Lantus-P-CN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC11681; U1111-1116-3661 (Other: UTN)
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin glargine (Experimental): injection once daily at bedtime
  Interventions: Drug: Insulin glargine (HOE901)
- NPH insulin (Active Comparator): injection once daily at bedtime or twice daily in the morning and at bedtime
  Interventions: Drug: NPH insulin

INTERVENTIONS:
Drug: Insulin glargine (HOE901) — Pharmaceutical form:aqueous solution for injection
  Route of administration: Subcutaneous
  Arms: Insulin glargine
Drug: NPH insulin — Pharmaceutical form:aqueous solution for injection
  Route of administration: Subcutaneous
  Arms: NPH insulin

SUMMARY:
Primary Objective:

6 To assess the efficacy of insulin glargine given once daily (QD) on glycosylated hemoglobin (HbA1c) levels over a period of 24 weeks in children with type 1 diabetes mellitus (T1DM) aged at least 6 years to less than 18 years.

Secondary Objectives:

* To assess the effects of insulin glargine compared to NPH insulin over 24 weeks on:

  * Percentage of patients reaching International Society of Pediatric and Adolescent Diabetes (ISPAD) recommended target of HbA1c < 7.5%,
  * Fasting blood glucose (FBG),
  * Nocturnal blood glucose (BG),
  * 24-hour blood glucose profile based on 8-point self-monitoring of blood glucose (SMBG) values,
  * Daily total insulin dose and basal insulin dose,
  * Rates of asymptomatic and/or symptomatic, severe, nocturnal and nocturnal symptomatic hypoglycemia.
* To assess the safety and tolerability of insulin glargine versus NPH insulin based on the occurrence of treatment-emergent adverse events (TEAEs).
* To assess anti-insulin and anti-glargine antibody development in both groups.
* To assess insulin glargine pharmacokinetic(PK) for all patients treated with insulin glargine in selected sites with approximately 45% of insulin glargine population to rule out accumulation tendency of insulin glargine after repeated dosing

DETAILED DESCRIPTION:
The study duration for each patient is 28 weeks +/- 7 day broken down as follows:

* Screening phase: up to 2 weeks
* Run-in phase: 1 week
* Treatment phase: 24 weeks
* Follow-up: 1 week

ELIGIBILITY:
Inclusion criteria:

- Paediatric patients diagnosed with T1DM aged at least 6 years to less than 18 years at screening.

Exclusion criteria:

* Treatment with oral or parenteral glucose-lowering medications other than insulin.
* HbA1c < 7% or > 12 % at screening.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2011-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Absolute change of glycosylated hemoglobin (HbA1c) | from baseline to week 24

SECONDARY OUTCOMES:
Percentage of patients reaching HbA1c < 7.5% | at week 24
Change in Fasting Blood Glucose (FBG) | from baseline to week 24
Change in nocturnal Blood Glucose (BG) | from baseline to week 24
Change in 24-hour blood glucose profile based on 8-point self-monitoring blood glucose (SMBG) | from baseline to week 24
Change in total insulin dose and basal insulin dose | from baseline to week 24
Rate of asymptomatic and/or symptomatic, severe, nocturnal, nocturnal symptomatic hypoglycemia. | during 24-week treatment period
Anti-glargine and anti-human insulin antibody assessment | at screening, week 4, week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (10):
- China (10):
  - Investigational Site Number 156006, Beijing
  - Investigational Site Number 156001, Beijing
  - Investigational Site Number 156007, Beijing
  - Investigational Site Number 156009, Changsha
  - Investigational Site Number 156008, Guangzhou
  - Investigational Site Number 156004, Hangzhou
  - Investigational Site Number 156016, Shanghai
  - Investigational Site Number 156005, Shanghai
  - Investigational Site Number 156019, Taiyuan
  - Investigational Site Number 156002, Wuhan

REFERENCES:
- [Derived] Liu M, Zhou Z, Yan J, Li P, Song W, Fu J, Chen X, Zhao W, Xi L, Luo X, Sha L, Deng X, Gong C. A randomised, open-labelstudy of insulin glargine or neutral protamine Hagedorn insulin in Chinese paediatric patients with type 1 diabetes mellitus. BMC Endocr Disord. 2016 Nov 26;16(1):67. doi: 10.1186/s12902-016-0146-2. PMID 27887605